CLINICAL TRIAL: NCT05784012
Title: Phase Ib/II Non-randomized Non-comparative Two-cohort Study of Niraparib and Dostarlimab Plus (Chemo)RadIotherapy in Locally-Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Two-cohort Study of Niraparib and Dostarlimab Plus (Chemo)RadIotherapy in Locally-Advanced Head and Neck Squamous Cell Carcinoma
Acronym: RADIAN
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Collaborators: GlaxoSmithKline (Industry); MFAR (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTCC-2022-01-RADIAN; 2023-000183-65 (EudraCT Number)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: non-metastatic; Oropharyngeal carcinoma; Laryngeal or hypopharyngeal carcinomas; Oral carcinoma; squamous cell carcinoma; radiotherapy; antiPD-1; PARP inhibitor
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Oropharyngeal Neoplasms; Laryngeal Diseases; Mouth Neoplasms; Carcinoma, Squamous Cell | interventions — dostarlimab; niraparib; Cisplatin; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Two cohorts:
  Cohort A: Patients who are candidates for definitive radiotherapy plus cisplatin (eligible for platinum).
  Cohort B: Patients who are ineligible for cisplatin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Three stages:
  Neoadjuvant: single dose of dostarlimab 500 mg intravenously on day -21 and niraparib 200 or 300 mg orally once daily starting on day -14 until 48 hours prior to the start of definitive radiotherapy (day 0).
  Concurrent: definitive radiotherapy (70 Gy in 35 fractions, 1 fraction per day from Monday to Friday) with concurrent Cisplatin at a dose of 100 mg/m2 intravenously on day 1 of week 1, week 4 and week 7.
  Maintenance: dostarlimab to be administered as a single infusion dose of 500 mg on day 1 every 21 days from week 11 to week 48. Niraparib will be given once daily at a dose of 200 or 300 mg in cycles of 21 days.
  Interventions: Drug: Dostarlimab; Drug: cisplatin plus radiotherapy; Drug: Niraparib
- Cohort B (Experimental): Three stages:
  Neoadjuvant: single dose of dostarlimab 500 mg intravenously on day -21 and niraparib 200 or 300 mg orally once daily starting on day -14 until the start of definitive radiotherapy (day 0).
  Concurrent: definitive radiotherapy (70 Gy in 35 fractions, 1 fraction per day from Monday to Friday). Niraparib is to be given once daily on a continous basis (200 to 300 mg), from w1 d1 until end of w10 in cycles of 21 days.
  Maintenance: dostarlimab to be administered as a single infusion dose of 500 mg on day 1 every 21 days from week 11 to week 48. Niraparib will be given once daily on a continous basis at a dose of 200 or 300 mg in cycles of 21 days.
  Interventions: Drug: Dostarlimab; Drug: Niraparib

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab 500 mg IV every 21 days in neoadjuvant and adjuvant stage.
Drug: Niraparib — Niraparib 200 or 300mg orally administered QD in neoadjuvant, concurrent with radiotherapy and adjuvant stage until completing week 48.
  Arms: Cohort B
Drug: cisplatin plus radiotherapy — In the concurrent phase
  Arms: Cohort A
Drug: Niraparib — Niraparib 200 or 300mg orally administered QD (Neoadjuvant and Maintenance stages).
  Arms: Cohort A

SUMMARY:
Multi-center, open-label, non-randomized, non-comparative two-cohort study for patients with locally-advanced squamous cell carcinoma arising from the larynx, hypopharynx, oropharynx (Stage III, IVA and IVB according to 8th TNM/AJCC ed.) and oral cavity (unresectable, stage IVB according to 8th TNM/ American Joint Committee on Cancer (AJCC) ed.) who are candidates for definitive radiotherapy plus cisplatin (Cohort A) or as single-modality (in cisplatin unfit patient population) (Cohort B) and will receive dostarlimab and niraparib in combination pre-, during and post- radiation.

Study has three parts:

1. Neoadjuvant phase (immune-conditioning phase): patients will receive 1 dose of dostarlimab + niraparib from day -14 prior to radiotherapy (up to 48h prior to radiotherapy (RT) in Cohort A and until RT in Cohort B).
2. Concurrent phase (radiosensitization): patients will receive definitive radiotherapy (70Gy in 35 fractions) with concurrent cisplatin (Cohort A) or with concurrent niraparib (Cohort B).
3. Maintenance: Following radiotherapy, patients will receive adjuvant dostarlimab plus niraparib until week 48 (37 cycles) in both cohorts.

ELIGIBILITY:
Inclusion Criteria:

Informed consent

1. Signed written and voluntary informed consent.
2. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
3. Age > 18 years, male or female.

   Disease characteristics
4. Have histologically confirmed new diagnosis of non-metastatic squamous cell carcinoma as assessed by the Investigator based on baseline imaging and clinical assessment that is either:

   1. Stage III HPV-related oropharyngeal carcinoma OR
   2. Stage III, IVA and IVB HPV-unrelated oropharyngeal, laryngeal or hypopharyngeal carcinomas. Stage IVB oral cavity squamous cell carcinomas may be eligible upon consultation with Sponsor if considered unresectable as per treating surgeon and multidisciplinary tumor board.

      * According to UICC/AJCC 8th Edition staging
5. Human papillomavirus (HPV)-relatedness in oropharyngeal primaries must be determined by positive p16 immunohistochemical staining on any tumor specimens and, if positive, confirmed by human papilloma virus (HPV) DNA testing by in situ hybridisation (ISH) or polymerase chain reaction (PCR). Positive p16 expression is defined as strong and diffuse nuclear and cytoplasmic staining in 70 % or more of the tumor cells. Local testing is acceptable.
6. Have an evaluable tumor burden assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI) based on RECIST 1.1 as assessed by the local site investigator/radiology.
7. Have provided newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for central biomarker analysis (fine needle aspirate (FNA) is not adequate).

   Repeat samples may be required if adequate tissue is not provided. Formalin-fixed, paraffin embedded tissue blocks are preferred to slides.

   Patient characteristics
8. Eastern cooperative oncology group (ECOG) performance status 0-1.
9. Patient must have adequate organ function as determined by the following:

   a. Hematology i. Absolute neutrophils > 1.5 x 109/L ii. Platelets > 100 x 109/L iii. Hemoglobin > 90 g/L b. Biochemistry i. Bilirubin < 1.5 x upper limit of normal (ULN) ii. aspartate aminotransferase (AST) and alanine transaminase (ALT) < 2.5 x ULN Note: Hematology test should be obtained without transfusion or receipt of colony stimulating factors within 4 weeks prior to obtaining sample.

   Specific criteria for Cohort A:

   iii. Creatinine clearance > 60 mL/min as per cockcroft -gault formula iv. Not presenting with peripheral neuropathy > grade 2 (CTCAE v5.0). v. Not presenting with clinically-significant hearing loss/tinnitus ≥ grade 3 (CTCAE v5.0).

   vi. 18-70 years old vii. Not presenting with cardiovascular disease: new york health association (NYHA) class II or higher, ischemic cardiovascular/cerebrovascular event in the past 12 months prior to inclusion in the study, clinically-significant peripheral arterial vasculopathy

   Specific criteria for Cohort B c. Patients considered unfit for cisplatin-based chemoradiotherapy, based on the following criteria (at least one): i. Creatinine clearance >30 but <60 mL/min ii. Impaired hearing loss/tinnitus ≥ grade 3 (CTCAE v5.0). iii. Peripheral neuropathy > grade 2 (CTCAE v5.0). iv. Age > 70 years old * Patients > 70 years old must be fit according to the G8 geriatric screening test (G8 > 14 points)
10. Evidence of post-menopausal status, or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
    2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Exclusion Criteria:

1. Early stages, defined as stage I-II according to Union for International Cancer Control (UICC) / American Joint Committee on Cancer (AJCC) 8th Edition staging in any localization, and including HPV-related and non-related.
2. Stage III-IVA oral cavity carcinoma considered resectable as per treating surgeon and/or multidisciplinary tumor board.
3. Has cancer outside of the oropharynx, larynx, and hypopharynx, nasopharyngeal, sinus, other para-nasal, or other unknown primary head and neck carcinoma (HNC).
4. Current history of other head and neck malignancies.
5. Any previous treatment for current head and neck cancer including systemic therapy, radiotherapy and/or surgery (except for a diagnostic biopsy) and no major surgery within 28 days prior to study treatment initiation.
6. Any previous radiation to the head and neck region that would result in overlap of fields for the current study.
7. Any previous radiotherapy treatment encompassing > 20 % of the bone marrow within 2 weeks or any radiotherapy within 1 week prior to Day 1 of protocol therapy.
8. Patients unable to swallow niraparib capsules/tablets.
9. Documented weight loss of >10 % during the last 4 weeks prior to study treatment initiation (unless adequate measures are undertaken for nutritional support), OR plasmatic albumin < 3.0 g/dL. No albumin transfusions are allowed within 2 weeks before study treatment initiation.
10. Active gastrointestinal bleeding, or any other uncontrolled bleeding requiring more than 2 red blood cell transfusions or 4 units of packed red blood cells within 4 weeks prior to study treatment initiation.
11. History of allergic or hypersensitivity reactions to any study drug or their excipients.
12. Patients with rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption should not take niraparib.
13. History of primary immunodeficiency, history of allogeneic organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of study treatment initiation or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy or grade ≥ 3 infusion reaction.
14. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease (e.g. colitis or Crohn's disease), diverticulitis with the exception of diverticulosis, celiac disease (controlled by diet alone) or other serious gastrointestinal chronic conditions associated with diarrhea), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome (granulomatosis with polyangiitis), rheumatoid arthritis, hypophysitis, uveitis, etc., within the past 3 years prior to the start of treatment. The following are exceptions to this criterion: vitiligo or alopecia; Patients with Grave's disease, vitiligo or psoriasis not requiring systemic treatment (within the last 2 years); Patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement. Any chronic skin condition that does not require systemic therapy.
15. History of interstitial lung disease e.g. pneumonitis requiring steroids (any dose) or immunomodulatory treatment within 90 days of planned start of the study therapy; or pulmonary fibrosis or evidence of pneumonitis on baseline CT scan.
16. Any concurrent chemotherapy, biologic, immunologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
17. Current or prior use of immunosuppressive medication within 14 days prior to starting dosing. The following are exceptions to these criteria:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection).
    2. Adrenal replacement steroid > 10 mg daily prednisone equivalent are permitted in the absence of active autoimmune disease.
    3. Steroids as premedication for hypersensitivity reactions (eg, computed tomography scan premedication).
18. Active or documented history of autoimmune disease within 2 years before screening, including:

    1. Active or prior documented inflammatory bowel disease (eg. Crohn's disease, ulcerative colitis).
    2. Patients with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, Grave's disease, Hashimoto's disease, or psoriasis not requiring systemic steroids and/or immunosuppressive agents within the past 2 years, are not excluded.
19. History of primary immune deficiency. History of stroke or transient ischemic attack within the previous 6 months.
20. History of uncontrolled hypertension: systolic BP >140 mmHg or diastolic BP >90 mmHg that has not been adequately treated or controlled prior to Day 1 of protocol therapy.
21. Any of the following cardiac abnormalities:

    1. Unstable angina pectoris,
    2. Congestive heart failure ≥ NYHA Class 2,
    3. QTc >480 milliseconds,
    4. Known Left ventricular ejection fraction (LVEF) < 50.
22. Concomitant medication known to cause prolonged QT that cannot be discontinued or changed to a different medication prior to enrollment.
23. History of organ transplant that requires use of immunosuppressive medications.
24. Patients with prior history of posterior reversible encephalopathy syndrome (PRES)
25. Known allergy or reaction to any components of niraparib and/or dostarlimab.
26. Subjects who are human immunodeficiency (HIV) positive.
27. Has a known history of or is positive for active hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (defined as hepatitis C virus (HCV) RNA [qualitative] is detected).

    1. hepatitis B virus (HBV) DNA must be undetectable and HBsAg negative at Screening Visit.
    2. Participants who have had definitive treatment for HCV are permitted if HCV RNA is undetectable at Screening Visit.
28. Female patients who are pregnant or breast-feeding.
29. Uncontrolled intercurrent illness including, but not limited to, ongoing or active clinically significant infection requiring parenteral antibiotics 2 weeks before treatment start, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events from niraparib and/or dostarlimab, or compromise the ability of the subject to give written informed consent.
30. Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study regimen or interpretation of patient safety or study results.
31. Any previous treatment with poly-ADP ribose polymerase (PARP), programmed death ligand (PD-L1) and/or cytotoxic T lymphocyte associated protein (CTLA-4) inhibitors.
32. History of another primary malignancy, except for:

    1. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study drug and of low potential risk for recurrence,
    2. Adequately treated non-melanoma skin cancer without evidence of disease,
    3. Adequately treated carcinoma in situ without evidence of disease.
33. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study medications.
34. Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1.
35. Any malabsorption problem that, in the investigator's opinion, would prevent adequate absorption of the study drug.
36. Known history of myelodysplastic syndrome (MDS) or a pre-treatment cytogenetic testing result at risk for a diagnosis of MDS/acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
1-year disease free survival | 1 year after the start of the study treatment
  Disease-free survival (DFS) is defined as the time from the date of study treatment initiation to the date of first record of any of the following events:
  Investigator determined:
  Locoregional progression or recurrence. Distant metastasis. Neck dissection or surgery performed for clinical or radiological disease progression (RECIST 1.1) > 20 weeks from the end of radiation therapy with tumor present on final pathology.
  Death due to any cause. Patients not presenting any of the previous events will be censored at the date of last assessment.

SECONDARY OUTCOMES:
Disease control rate | Throughout the study period, approximately 36 months
  Disease Control Rate (DCR) is defined as the percentage of patients who have achieved complete response, partial response and stable disease by RECIST 1.1 at a certain time point. DCR will be evaluated at 12, 18 and 24 and 36 months.
Locoregional control | Throughout the study period, approximately 36 months
  Time to locoregional failure is defined as the time from the date of study treatment initiation to the date of the first record of appearance of local or regional progression/recurrence, to the date of neck dissection > 20 weeks performed for clinical or radiological (RECIST 1.1) disease progression from the end of radiation therapy with tumor present, or to the date of surgery of primary tumor with tumor present performed for clinical or radiological (RECIST 1.1) disease progression, whichever comes first.
Distant control | Throughout the study period, approximately 36 months
  Time to distant metastasis is defined as the time from the date of study treatment initiation to the date of first record of appearance of distant metastasis. Locoregional failure or second cancers diagnosed before the distant metastases are not considered events of interest for this endpoint.
Event-free survival | Throughout the study period, approximately 36 months
  Event-free survival (EFS) is defined as the time from the date of study treatment initiation to the date of first record of any of the following events:
  Investigator determined:
  Locoregional progression or recurrence. Distant metastasis.
  Surgery:
  Surgery for persistent or residual disease at the primary tumor site with tumor present on final pathology.
  Neck dissection or surgery performed for clinical or radiological disease progression (RECIST 1.1) > 20 weeks from the end of radiation therapy with tumor present on final pathology.
  Death due to any cause. Patients not presenting any of the previous events will be censored at the date of last assessment.
Overall survival | Throughout the study period, approximately 36 months
  Event-free survival (EFS) is defined as the time from the date of study treatment initiation to the date of first record of any of the following events:
  Investigator determined:
  Locoregional progression or recurrence. Distant metastasis.
  Surgery:
  Surgery for persistent or residual disease at the primary tumor site with tumor present on final pathology.
  Neck dissection or surgery performed for clinical or radiological disease progression (RECIST 1.1) > 20 weeks from the end of radiation therapy with tumor present on final pathology.
  Death due to any cause. Patients not presenting any of the previous events will be censored at the date of last assessment.
Frequency of treatment-related adverse events | Throughout the study period, approximately 36 months
  Number of patient who experienced treatment-related adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Oliva, M.D., Study Chair — Institut Català D´Oncologia (ICO) Hospitalet de Llobregat; Ricard Mesia, M.D. Ph.D., Study Chair — Institut Català d''Oncologia (ICO) Badalona
Locations (5):
- Spain (5):
  - Institut Catalá d'Oncologia (ICO) BADALONA, Badalona, Catalonia
  - Hospital Universitario Valle Hebron, Barcelona, Catalonia
  - Hospital Clinic de Barcelona, Barcelona, Catalonia
  - Institut Catalá d'Oncologia (ICO) Hospitalet, L'Hospitalet de Llobregat, Catalonia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: No